CLINICAL TRIAL: NCT05245474
Title: Efficacy and Safety of Neoadjuvant Long-course Chemoradiation Plus Tislelizumab in Mid-low Locally Advanced Rectal Cancer: a Phase II, Multi-center, Open-label, Randomized Controlled Trial (POLARSTAR Trial)
Brief Title: Neoadjuvant Long-course Chemoradiation Plus PD-1 Blockade for Mid-low Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Xuanwu Hospital, Beijing (Other); Beijing Hospital (Other Government); Peking Union Medical College Hospital (Other); Peking University First Hospital (Other); Peking University People's Hospital (Other); Peking University Cancer Hospital & Institute (Other); BeiGene (Industry)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFH-POLARSTAR
Record Dates: First submitted 2022-02-06; First posted 2022-02-18 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: LARC; radiation; chemoradiation; PD-1; Tislelizumab; neoadjuvant; randomized; controlled
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Masking Description: Masking is not practically possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRT+concurrent PD-1 inhibition (Experiment Arm 1) (Experimental): Long-course chemoradiation plus PD-1 inhibition (Tislelizumab 200mg, 3 times, 3-week interval) starting on Day 8 of radiation therapy. TME surgery is scheduled in 8~12 weeks after completion of radiation.
  Interventions: Combination Product: Long-course chemoradiation, with or without Tislelizumab (PD-1 inhibitor)
- CRT+sequential PD-1 inhibition (Experiment Arm 2) (Experimental): Long-course chemoradiation plus PD-1 inhibition (Tislelizumab 200mg, 3 times, 3-week interval) starting on Day 15 after completion of radiation therapy. TME surgery is scheduled in 8~12 weeks after completion of radiation.
  Interventions: Combination Product: Long-course chemoradiation, with or without Tislelizumab (PD-1 inhibitor)
- CRT without PD-1 inhibition (Control Arm) (Active Comparator): Long-course chemoradiation plus PD-1 inhibition with no PD-1 inhibition. TME surgery is scheduled in 6~12 weeks after completion of radiation.
  Interventions: Combination Product: Long-course chemoradiation, with or without Tislelizumab (PD-1 inhibitor)

INTERVENTIONS:
Combination Product: Long-course chemoradiation, with or without Tislelizumab (PD-1 inhibitor) — Tislelizumab is added to long-course chemoradiation (CRT) of LARC patients, with CRT+concurrent Tislelizumab for Arm 1, CRT+sequential Tislelizumab for Arm 2, and CRT only for Arm 3

SUMMARY:
This is a phase II/III, multi-center, open-label, 3-arm, randomized controlled trial assessing the efficacy and safety of neoadjuvant long-course chemoradiation combined with Tislelizumab (PD-1 inhibitor) and subsequent TME surgery, by comparing assorted endpoints between two experiment groups (Experiment group 1: chemoradiation+concurrent PD-1 inhibitor; Experiment group 2: chemoradiation+sequential PD-1 inhibitor) with a control group (chemoradiation only).

DETAILED DESCRIPTION:
This phase II, multi-center, open-label, 3-arm, randomized trial aims to recruit patients aged 18-75 years, diagnosed histologically as rectal adenocarcinoma, without metastasis (by CT), staged II/III (by MRI, T4b excluded), with distal margin within 10cm to anal verge. All patients should have no history of immune diseases, nor history of immunotherapy or radiotherapy. Sample size was thoroughly calculated to be 186. Eligible participants will be randomly assigned to Experiment Arm 1 (50.4Gy radiation, capecitabine, and anti-PD1 starting at Day 8 of radiation), Experiment Arm 2 (50.4Gy radiation, capecitabine, and anti-PD1 starting 2 weeks after completion of radiation), and Control Arm (50.4Gy radiation, capecitabine) in a 1:1:1 ratio. Randomization is stratified by different centers, with a block size of 6. For both experiment arms, Tislelizumab (anti-PD1) is scheduled to be administered at 200mg each time for 3 times, with 3-week intervals. The primary endpoint is pCR rate, and secondary endpoints include sphincter-preserving rate, adverse event rates, and DFS and OS rate at 2, 3 and 5 years post-operation. Data will be analyzed with an intention-to-treat or modified intention-to-treat approach.

ELIGIBILITY:
Inclusion Criteria:

* aged 18~75
* ECOG score 0~2
* biopsy diagnosed rectal adenocarcinoma, distal margin within 10cm to anal verge
* no distant metastasis, staged II/III (T4b excluded) by MRI
* maximum diameter of rectal cancer lesion≥10mm according to baseline CT or MRI (i.e. a "measurable lesion" as per RECIST 1.1 criteria)
* willing and able to comply with study protocol
* consent to the use of blood and tissue specimens for study
* no history of previous anti-tumor treatment (e.g. radiation, chemo, immuno, bio, herbal, etc.)
* no disorders/diseases of immune system (e.g. systemic lupus erythematosus, rheumatoid arthritis, systemic vasculitis, scleroderma, pemphigus, dermatomyositis, mixed connective tissue disease, autoimmune hemolytic anemia, hyperthyroidism/hypothyroidism, ulcerative colitis, autoimmune hemolytic anemia, HIV infection, etc.)
* no significant dysfunction of major viscera (e.g. heart, lung, liver, kidney, etc.)
* no jaundice or gastrointestinal obstruction
* no acute/ongoing infection
* no significant irregularities in blood routine test and biochemical test results, particular requirements include: neutrophils≥1.5×109/L, HGB≥80g/L, platelet≥100×109/L, serum creatinine≤1.5×ULN, total bilirubin≤1.5×ULN, ALT、AST≤2.5×ULN
* no social or mental disorder
* for women of child-bearing age, a negative result of serological pregnancy test is required, and effective contraception measures from inclusion till 60 days after the last dose of study drug is required

Exclusion Criteria:

* multiple cancers, or with concomitant malignant tumors besides rectal cancer
* having received any anti-cancer treatment (surgery, drugs, etc.) in the past 5 years
* history of recent major surgery
* with condition that affects the absorption of capecitabine via gastrointestinal tract (e.g. inability to swallow, nausea, vomiting, chronic diarrhea, etc.)
* with uncontrolled, severe, concomitant diseases of any sort
* allergic to any of the ingredients under study
* estimated survival ≤ 5 years due to any reason
* preparing for or having previously received organ or bone marrow transplant
* having received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to inclusion
* for patients with history of disorder of central nervous system, investigator discretion is required as to whether the clinical severity prevents the signing of informed consent or affects the patient's oral medication compliance
* with other conditions/issues that may affect the study results or cause the study treatment to be terminated halfway (e.g. alcoholism, drug abuse, etc.)
* pregnant or lactating women, or women intending on conception during treatment period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | within 10 days after surgery
  pathological complete response rate

SECONDARY OUTCOMES:
NAR score | within 10 days after surgery
  neoadjuvant rectal score
2-y OS rate | 2 year
  2-year overall survival rate
2-y DFS rate | 2 year
  2-year disease free survival rate
3-y OS rate | 3 year
  3-year overall survival rate
3-y DFS rate | 3 year
  3-year disease free survival rate
5-y OS rate | 5 year
  5-year overall survival rate
5-y DFS rate | 5 year
  5-year disease free survival rate
median OS time | 0~60 months
  median length (in months) of overall survival period
median DFS time | 0~60 months
  median length (in months) of disease free survival period
R0 resection rate | within 10 days after surgery
  rate of R0 resection
sphincter preserving rate | instantly after surgery
  proportion of patients with preserved anal sphincter
nearly pCR rate | within 10 days after surgery
  nearly pathological complete response rate
ORR | before surgery
  objective response rate
immune-related adverse event rate | from commencing of PD-1 inhibition to the 30th day after surgery
  adverse event rate that is deemed to be associated with PD-1 inhibition
Grade 3+ immune-related adverse event rate | from commencing of PD-1 inhibition to the 30th day after surgery
  adverse event (above Grade 3) rate that is deemed to be associated with PD-1 inhibition
treatment-related adverse event rate | from commencing of treatment to the 30th day after surgery
  adverse event rate that is deemed to be associated with all treatments
Grade 3+ treatment-related adverse event rate | from commencing of treatment to the 30th day after surgery
  adverse event (above Grade 3) rate that is deemed to be associated with all treatments
cCR rate | before surgery
  clinical complete response rate
incidence rate of surgical complications | within 30 days after surgery
  incidence rate of surgical complications within 30 days after surgery
incidence rate of Grade 3+ surgical complications | within 30 days after surgery
  incidence rate of Grade 3+ surgical complications within 30 days after surgery
quality of life score | during the 5 years after surgery
  quality of life score during the 5 years after surgery, multiple timepoint assessment

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Principal Investigator — Beijing Friendship Hospital
Locations (8):
- China (8):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No
Export of individual patient data is a sensitive issue according to current Chinese laws

REFERENCES:
- [Background] Pang K, Yang Y, Zhao P, Wu G, Li J, Gao J, Yao H, Yang Y, Zhang Z. Adding immune checkpoint blockade to neoadjuvant chemoradiation in locally advanced rectal cancer. Br J Surg. 2022 Oct 14;109(11):1178-1179. doi: 10.1093/bjs/znac298. No abstract available. PMID 36001602
- [Derived] Pang K, Sun P, Liu X, Yang D, Zhao P, Huang Y, Cao S, Gao Y, Chen G, Yu H, Duan L, Yang Y, Zhang Z. Development of the rationale of a personalized cancer vaccine based on the in situ vaccine effect of radiotherapy: a mechanistic study of the POLARSTAR trial. Cancer Immunol Immunother. 2025 Nov 12;74(12):369. doi: 10.1007/s00262-025-04229-3. PMID 41222702
- [Derived] Yang Y, Pang K, Lin G, Liu X, Gao J, Zhou J, Xu L, Gao Z, Wu Y, Li A, Han J, Wu G, Wang X, Li F, Ye Y, Zhang J, Chen G, Wang H, Kong Y, Wu A, Xiao Y, Yao H, Zhang Z. Neoadjuvant chemoradiation with or without PD-1 blockade in locally advanced rectal cancer: a randomized phase 2 trial. Nat Med. 2025 Feb;31(2):449-456. doi: 10.1038/s41591-024-03360-5. Epub 2025 Jan 6. PMID 39762418
- [Derived] Pang K, Yang Y, Tian D, Zeng N, Cao S, Ling S, Gao J, Zhao P, Wang H, Kong Y, Zhang J, Chen G, Deng W, Bai Z, Jin L, Wu G, Zhu D, Wang Y, Zhou J, Wu B, Lin G, Xiao Y, Gao Z, Ye Y, Wang X, Li A, Han J, Yao H, Yang Y, Zhang Z. Long-course chemoradiation plus concurrent/sequential PD-1 blockade as neoadjuvant treatment for MMR-status-unscreened locally advanced rectal cancer: protocol of a multicentre, phase 2, randomised controlled trial (the POLAR-STAR trial). BMJ Open. 2023 Sep 12;13(9):e069499. doi: 10.1136/bmjopen-2022-069499. PMID 37699634
- See also: Study protocol was published as an abstract on 2022 ESMO Congress — https://doi.org/10.1016/j.annonc.2022.07.1868